CLINICAL TRIAL: NCT05894603
Title: Post-marketing Surveillance Study of the Effectiveness and Safety of New Oral Antivirals for Outpatients With Mild-moderate COVID-19
Brief Title: Effectiveness and Safety of New Oral Antivirals for COVID-19
Acronym: ESOA-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Other Study IDs: ESOA-19; EUPAS48186 (Other: EU PAS Register - ENCePP)
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Post-marketing surveillance; COVID-19; Antivirals; Effectiveness; Safety
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination; molnupiravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral antiviral A: Patients with an indication for treatment with nirmatrelvir + ritonavir (Paxlovid®).
  Interventions: Drug: Nirmatrelvir/ritonavir
- Oral antiviral B: Patients with an indication for treatment with molnupiravir (Lagevrio®).
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — Nirmatrelvir/ritonavir
  Other Names: Paxlovid
  Groups: Oral antiviral A
Drug: Molnupiravir — Molnupiravir
  Other Names: Lagevrio
  Groups: Oral antiviral B

SUMMARY:
There is an increased lack of short- and long-term real-life effectiveness and safety data on new oral antivirals authorised and commercialised to treat COVID-19. To date, only two clinical trials have been published with data on the efficacy and safety of the use of the Paxlovid® and Lagevrio®. Since there is a public health, political, social and economic pressure to prevent severity, hospitalisation and death from COVID-19, monitoring the effectiveness and safety of commercialised oral antiviral therapies against COVID-19 has become emergent pharmacovigilance and public health task. The objective of the study is to monitor the post-marketing safety and effectiveness of the new oral antivirals indicated for the treatment of COVID-19, namely Nirmatrelvir/Ritonavir (Paxlovid®) and Molnupiravir (Lagevrio®), having as holders of the Authorization of Market introduction to Pfizer Europe MA EEIG and Merck Sharp & Dohme B.V., respectively.

DETAILED DESCRIPTION:
There is an increased lack of short- and long-term real-life effectiveness and safety data on new oral antivirals authorised and commercialised to treat COVID-19. To date, only two clinical trials have been published with data on the efficacy and safety of the use of the Paxlovid® and Lagevrio®. Since there is a public health, political, social and economic pressure to prevent severity, hospitalisation and death from COVID-19, monitoring the effectiveness and safety of commercialised oral antiviral therapies against COVID-19 has become emergent pharmacovigilance and public health task6.

A real-life cohort event monitoring system allows for the monitoring of newly introduced oral antivirals, in addition to existing spontaneous reporting systems and healthcare database studies (i.e., secondary data), as it is complementary to these systems in several ways. First, it is better suited to capture the more frequent AE, including those that are not medically attended. It generates more comprehensive safety data, e.g. on disease course and the impact of the AE. Moreover, there is insufficient data on these new medicines in real clinical practice, particularly from large-scale studies on the long-term efficacy or safety.

This work, with scientific and academic interest but, essentially, clinical and regulatory importance, constitutes a duty of the regional pharmacovigilance units. As such, it is also an obligation of the Pharmacy and Therapeutics Commissions, based on the legislation in force, to "collaborate in studies to monitor the safety and effectiveness of medicines promoted in the context of the National Pharmacovigilance System".

ELIGIBILITY:
Inclusion Criteria:

Participants eligible to be included in the study are identified by medical prescribing of one of the drugs under study, and either the medicine recipient or their proxy should:

1. Comply with the eligibility criteria for prescribing these drugs (including patients ≥ 18 years old), according to Norm nr 005/2022 of the General Directorate of Health of Portugal*;
2. Enrol in the study within the first 72 hours after dispensing treatment;
3. Be able to understand the Portuguese language;
4. Available for follow-up during study time;
5. Provide informed consent.

   * Compliance with the eligibility criteria for prescribing these drugs is the sole responsibility of the prescriber who assesses the patient, so the study centres only include patients referred by the prescriber.

Exclusion Criteria:

Will be considered ineligible participants those who:

1. Are not available for follow-up and monitoring;
2. Participate in phase I, II, III or IV clinical trials;
3. Life expectancy is less than one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving the oral antivirals against COVID-19 - Paxlovid® or Lagevrio®.
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | 6 days after onset treatment for both drugs.
  The incidence of AE (with particular focus on AE of special interest) that emerge during or after the treatment period, serious AE, and AE leading to discontinuation of the treatment, as coded according to the MedDRA. Incidence data will be provided for each treatment group within the safety analysis population, including all patients who received at least one drug dose.
  The occurrence of AE will be asked in open question / unsolicited. For each reported AE, date of onset, outcome, duration of symptoms (if recovered), and severity/impact of the symptoms (including medical assistance & hospitalisation) will be asked.
Safety outcome | 39 days after treatment onset for nirmatrelvir/ritonavir cohort.
  The incidence of AE (with particular focus on AE of special interest) that emerge during or after the treatment period, serious AE, and AE leading to discontinuation of the treatment, as coded according to the MedDRA. Incidence data will be provided for each treatment group within the safety analysis population, including all patients who received at least one drug dose.
  The occurrence of AE will be asked in open question / unsolicited. For each reported AE, date of onset, outcome, duration of symptoms (if recovered), and severity/impact of the symptoms (including medical assistance & hospitalisation) will be asked.
Safety outcome | 19 days after treatment onset for molnupiravir cohort.
  The incidence of AE (with particular focus on AE of special interest) that emerge during or after the treatment period, serious AE, and AE leading to discontinuation of the treatment, as coded according to the MedDRA. Incidence data will be provided for each treatment group within the safety analysis population, including all patients who received at least one drug dose.
  The occurrence of AE will be asked in open question / unsolicited. For each reported AE, date of onset, outcome, duration of symptoms (if recovered), and severity/impact of the symptoms (including medical assistance & hospitalisation) will be asked.
Effectiveness outcome | 29 days after treatment onset for both drugs.
  The incidence of hospitalisation for any cause (defined as ≥24 hours of acute care in a hospital or any similar facility) or death for any cause through day 29.

SECONDARY OUTCOMES:
Adherence to treatment | 6 days after onset treatment for both drugs.
  Will be measured using the self-reported 7-item Measure Treatment Adherence (MTA) tool validated for the Portuguese Population. The MTA is a psychometric tool derived from the Morisky et al. questionnaire and evaluates the individuals' behaviour concerning the daily use of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Junqueira Polónia, MD, PhD, Study Director — Universidade do Porto
Locations (6):
- Portugal (6):
  - Hospital do Divino Espírito Santo de Ponta Delgada, EPE, Açores
  - Centro Hospitalar de Lisboa Ocidental, EPE, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Porto
  - Centro Hospitalar e Universitário de São João, EPE, Porto
  - Centro Hospitalar Universitário de Santo António, EPE, Porto
  - Unidade de Saúde Familiar - Homem do Leme (ACES Porto Ocidental), Porto